CLINICAL TRIAL: NCT02712385
Title: Stroke Prevention Rehabilitation Intervention Trial of Exercise - SPRITE - A Feasibility and Pilot Study
Brief Title: Stroke Prevention Rehabilitation Intervention Trial of Exercise (SPRITE)
Acronym: SPRITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Prof Frank Kee, Professor of Public Health, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDV/5053/14
Record Dates: First submitted 2016-02-28; First posted 2016-03-18 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Cerebrovascular Disorders
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: The intervention groups will be getting access to a home-based rehabilitation, 'The Healthy Brain Rehabilitation Manual', telephone follow-up with either a GP or stroke nurse and a pedometer.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control - usual care (No Intervention): Usual post-TIA/minor stroke care as per current healthcare system protocol will be given to patients in control group and details will be recorded.
- Manual (Active Comparator): Receiving usual post-TIA/minor stroke care plus 'The Healthy Brain Rehabilitation Manual'.
  Interventions: Other: 'The Healthy Brain Rehabilitation Manual'; Procedure: Usual care
- Manual + pedometer, 1 (Active Comparator): Receiving usual post-TIA/minor stroke care plus 'The Healthy Brain Rehabilitation Manual' and a pedometer with telephone follow-up from a General Practitioner.
  Interventions: Other: 'The Healthy Brain Rehabilitation Manual'; Device: Pedometer; Procedure: Usual care; Behavioral: Telephone follow-up
- Manual + pedometer, 2 (Active Comparator): Receiving usual post-TIA/minor stroke care plus 'The Healthy Brain Rehabilitation Manual' and a pedometer with telephone follow-up from a Stroke nurse.
  Interventions: Other: 'The Healthy Brain Rehabilitation Manual'; Device: Pedometer; Procedure: Usual care; Behavioral: Telephone follow-up

INTERVENTIONS:
Other: 'The Healthy Brain Rehabilitation Manual' — The Healthy Brain Rehabilitation Manual is a home-based rehabilitation manual developed for the post-TIA and minor stroke population caused by ischaemic events. The manual addresses all the secondary prevention factors required post-ischaemic TIA/minor stroke, e.g. smoking cessation, physical activity promotion.
  Arms: Manual; Manual + pedometer, 1; Manual + pedometer, 2
Device: Pedometer — Pedometer used to measure step counts as an objective measurement of level of physical activity.
  Arms: Manual + pedometer, 1; Manual + pedometer, 2
Procedure: Usual care — Usual care provided by healthcare system for patients who suffer a TIA or minor stroke will be recorded and form 'active comparator' control.
  Arms: Manual; Manual + pedometer, 1; Manual + pedometer, 2
Behavioral: Telephone follow-up — Telephone follow-up by either a General Practitioner (GP) or Stroke nurse.
  Arms: Manual + pedometer, 1; Manual + pedometer, 2

SUMMARY:
BACKGROUND - Approximately 1,700 transient ischaemic attacks (TIAs) occur annually in NI with TIA survivors often being left with considerable functional impairment. TIA and strokes share common risk factors with cardiovascular disease. Cardiac rehabilitation post-myocardial infarction has shown significant reductions in morbidity and mortality, with home-based programmes producing better adherence and similar outcomes to hospital-and community-based programmes. However, the value of rehabilitation programmes for stroke prevention following a TIA or minor stroke is unclear.

AIMS - to determine if a novel rehabilitation programme, 'The Healthy Brain Rehabilitation Manual', for TIA/minor stroke patients can be developed, using MRC guidelines for developing complex health service interventions, from an approved home-based cardiac rehabilitation programme (the 'Heart Manual') and to undertake feasibility and pilot studies of the novel programme.

METHODS-All patients attending a TIA clinic in Belfast within 4 weeks of their first TIA/mild stroke will be invited to participate. The novel home-based programme manual will be developed following systematic reviews of the literature and qualitative exploration with the target population, using focus groups. A feasibility study will initially be undertaken lasting 6 weeks and then developed into a pilot trial of 12 weeks duration. The feasibility will recruit to 3 different treatments: (1) standard care; (2) standard care plus the manual; (3) standard care, manual plus a pedometer. Whilst for the pilot study there will also be 3 arms but this will include: 1) control group; 2) manual and pedometer supported by telephone follow-up with a GP; 3) manual and pedometer supported by telephone follow-up with a stroke nurse. Interviews and focus groups will be employed to assess the interventions' acceptability. The intervention, 'The Healthy Brain Rehabilitation Manual' will be refined and modified at all stages of the research.

CONCLUSIONS - The findings will inform the development of a novel secondary prevention programme, 'The Healthy Brain Rehabilitation Manual', for TIA/minor stroke patients and of a trial to test its effectiveness and longer-term potential to improve outcomes for TIA/stroke patients.

DETAILED DESCRIPTION:
METHODS - The development of the novel home-based rehabilitation programme, adapted from the "Heart Manual", will follow the guidelines of the MRC for developing complex health service interventions. The steps of the guidelines include: 1) exploring relevant theory; 2) modelling the preliminary intervention by selecting the main components based on the literature and qualitative research; 3) pilot-testing the preliminary intervention; 4) developing the definitive randomised controlled trial; and, 5) implementing and evaluating the randomised controlled trial over the long-term. This study focuses on the first three steps of the MRC framework.

Exploration of relevant theory - Initially, literature relating to cardiac rehabilitation and secondary prevention of TIAs and minor stroke will be reviewed following searches in appropriate databases with input from a medical librarian. The research team (including the applicant, supervisors, collaborators and steering group) will discuss key findings and identify those deemed appropriate to the study setting, with identification of appropriate behaviour change theory using behaviour change taxonomy.

Recruitment: Participants will be recruited from one TIA/ 'minor' stroke assessment unit, based in the Ulster Hospital for the feasibility study and from 4 sites for the pilot study (Royal Victoria Hospital, Ulster Hospital, Antrim and Craigavon Area Hospitals). Patients are typically seen within one week of suffering neurological symptoms suggestive of TIA. After confirmation of diagnosis and initial management on the day of presentation, the attending physician will offer patients a study information sheet and an invitation to participate. If the patient agrees to being contacted, the researcher will telephone twenty-four hours later to invite them to attend the Clinical Research Facility, QUB to participate in the study and written, informed consent will be obtained. The numbers of those who decline to participate in the study will be recorded to provide information about recruitment rates.

Developing the intervention: From those who agree to participate, an initial purposeful sample of patients will be invited to focus groups. Participants will be given the manual approximately a week before the focus group and asked to read it before attending the focus group. The topic guide for focus groups will be based on findings from the literature review and will include the formatting and lay-out of the manual, manual content and potential improvements to the manual. Health and social care staff involved in the clinical care of TIA and stroke patients, members of voluntary organisations, relatives and carers will also be invited to participate in a focus group: initial plans are that a sample of these individuals would be invited to a single group. Participants' and professionals' experiences of and attitudes towards key interventions identified from the literature will also be used in modelling the pilot intervention. With each participant's consent, interviews and focus groups will be audio-recorded and transcribed. Two researchers will then analyse the transcripts independently by: familiarisation; identifying a thematic framework; indexing; charting; and, mapping and interpretation.

Feasibility and then pilot study of the intervention - Baseline assessment: Following analysis of the findings of the literature review and qualitative data, the home-based vascular rehabilitation manual will be developed, adapting the "Heart Manual" (now referred to as 'The Healthy Brain Rehabilitation Manual') accordingly. We plan to conduct both a feasibility and pilot studies of our intervention. As described above, prospective trial participants will be invited to attend the Clinical Research Facility within 4 weeks of their initial TIA/'minor' stroke event, for initial assessment, at which their written consent to participate will be sought. Baseline assessments (taking approximately 60 minutes) will be completed prior to randomisation to ensure allocation concealment. All patients will initially undertake a sub maximal exercise test under the supervision of a trained physician. For the pilot study, all will be given, with appropriate instructions, an accelerometer to wear for one week to provide a blinded baseline physical activity assessment and these will be returned to the applicant after one week.

Randomisation: Block randomisation will be used and patients will be stratified, based on age, sex and diagnosis (TIA/'minor' stroke). Study group allocation will be revealed to participants only at the end of the baseline assessment and following completion of all initial measurements (except accelerometry).

Interventions: The feasibility will recruit to 3 different treatments: (1) standard care; (2) standard care plus the manual; (3) standard care, manual plus a pedometer. Whilst for the pilot study there will also be 3 arms but this will include: 1) control group; 2) manual and pedometer supported by telephone follow-up with a GP; 3) manual and pedometer supported by telephone follow-up with a stroke nurse. The control group (Group 1) will follow standard care guidelines as per treatment protocols and provided by their healthcare professionals at the hospital clinic. 'The Healthy Brain Rehabilitation Manual' programme will be explained to the appropriate participants by the applicant at the end of the baseline assessment. The use of the pedometer, an approach to its use in goal setting and an accompanying diary will also be explained to the relevant participants at that time.

'The Healthy Brain Rehabilitation Manual' will address each of the modifiable vascular risk factors, managing one risk factor each week, whilst encouraging the patient to slowly increase their activity over the (proposed) six week programme in the setting of their home and addressing the issues of anxiety and depression following the diagnosis of TIA or 'minor' stroke. The manual therefore involves education and motivation of the patient to address these risk factors. The facilitator (the applicant (a General Practitioner) and/or a stroke nurse) will also help them identify local support resources, for example smoking cessation services, through telephone contact. 'The Healthy Brain Rehabilitation Manual' will utilise the behaviour change techniques of goal setting, barrier identification, setting graded tasks, self monitoring, feedback, relapse prevention and stress management. Self-set pedometer targets will emerge during discussion with the facilitator who will use simple motivational interviewing techniques and advise keeping a daily step-count diary. Telephone follow-up review, with the applicant, will take place at one and four weeks as per usual "Heart Manual" care for the feasibility study as well as at eight weeks for the pilot study, unless the findings of initial qualitative work would suggest that an alternative design of a follow-up plan would be appropriate. These reviews will include advice regarding addressing the modifiable vascular risk factors and, if appropriate, issues with the home-based vascular rehabilitation programme ('The Healthy Brain Manual') and pedometer targets.

Review assessment: All participants will have a 6 week (feasibility study) and a 3 month (pilot study) follow-up review appointment. This review should take approximately sixty minutes to complete. For the pilot study, all participants will be asked to wear an accelerometer again, for one week, to provide a post-intervention physical activity assessment and to return this to the researcher following this period.

End-of study qualitative assessment: At the end of the pilot study, all participants will be asked about their perceptions of the relevance, acceptability and value of the intervention, using different qualitative techniques, including questionnaires, focus groups and/or semi structured interviews.

The manual will be developed at all stages of the research process as per the MRC guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* male or female
* attendee at a participating TIA clinic within 4 weeks of a first suspected TIA
* diagnosed with a TIA or 'minor' stroke, due to atherosclerosis or small vessel occlusion (diagnosis based on the TOAST classification system (69)(70), following neurological examination and neuroimaging (32)).

Exclusion Criteria:

* patients who have experienced more than one TIA and/or stroke
* inability to give informed consent
* presenting after 4 weeks of their first suspected TIA and/or 'minor' stroke
* contra-indication for exercise training, based on guidelines of the American College of Sports Medicine(72)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment to the studies | 12 weeks (pilot study)
  Recruitment rate calculated as percentage of potentially eligible patients who agree to participate

SECONDARY OUTCOMES:
Change in Level of physical activity | Baseline to 12 weeks
  Physical activity measured as step count (steps/day) assessed at baseline and 12 weeks, to determine extent of change. Also accelerometer data over the same timeframe.
Change in Body Mass Index (BMI) | Baseline to 12 weeks
  BMI measured at baseline and 12 weeks, to determine extent of change
Change in Quality of life | Baseline to 12 weeks
  Quality of life assessed at baseline and 12 weeks, to determine extent of change
Change in Blood pressure | Baseline and 12 weeks
  Systolic and diastolic blood pressure measured at baseline and 12 weeks.
Change in Physical function | Baseline and 12 weeks
  Distance walked in two minutes assessed by the two minute walk test at baseline and 2 weeks to determine extent of change in measurement

CONTACTS AND LOCATIONS:
Overall Officials: Frank Kee, MRCGP, MD, Principal Investigator — Queen's University, Belfast
Locations (4):
- United Kingdom (4):
  - Ulster Hospital, Belfast, Antrim
  - Royal Group of Hospitals, Belfast, Antrim
  - Craigavon Area Hospital, Craigavon, Armagh
  - Antrim Area, Antrim

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available

REFERENCES:
- [Background] Heron N, Kee F, Donnelly M, Tully MA, Cupples ME. Systematic review of the use of behaviour change techniques (BCTs) in home-based cardiac rehabilitation programmes for patients with cardiovascular disease--protocol. Syst Rev. 2015 Nov 17;4:164. doi: 10.1186/s13643-015-0149-5. PMID 26577666
- [Background] Heron N, Kee F, Donnelly M, Cupples ME. Systematic review of rehabilitation programmes initiated within 90 days of a transient ischaemic attack or 'minor' stroke: a protocol. BMJ Open. 2015 Jun 18;5(6):e007849. doi: 10.1136/bmjopen-2015-007849. PMID 26088808
- [Background] Heron N, Kee F, Cardwell C, Tully MA, Donnelly M, Cupples ME. Secondary prevention lifestyle interventions initiated within 90 days after TIA or 'minor' stroke: a systematic review and meta-analysis of rehabilitation programmes. Br J Gen Pract. 2017 Jan;67(654):e57-e66. doi: 10.3399/bjgp16X688369. Epub 2016 Dec 5. PMID 27919935
- [Background] Cupples M, Heron N. What to do after cardiac rehabilitation programs: the role of the general practitioner in cardiovascular prevention. Monaldi Arch Chest Dis. 2016 Oct 14;86(1-2):755. doi: 10.4081/monaldi.2016.755. PMID 27748471
- [Background] Heron N, Kee F, Donnelly M, Cardwell C, Tully MA, Cupples ME. Behaviour change techniques in home-based cardiac rehabilitation: a systematic review. Br J Gen Pract. 2016 Oct;66(651):e747-57. doi: 10.3399/bjgp16X686617. Epub 2016 Aug 1. PMID 27481858
- [Result] Heron N, Kee F, Mant J, Reilly PM, Cupples M, Tully M, Donnelly M. Stroke Prevention Rehabilitation Intervention Trial of Exercise (SPRITE) - a randomised feasibility study. BMC Cardiovasc Disord. 2017 Dec 12;17(1):290. doi: 10.1186/s12872-017-0717-9. PMID 29233087
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251
- [Derived] Heron N. Optimising secondary prevention in the acute period following a TIA of ischaemic origin. BMJ Open Sport Exerc Med. 2017 Jan 6;2(1):e000161. doi: 10.1136/bmjsem-2016-000161. eCollection 2016. PMID 29616144

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT02712385/SAP_000.pdf